CLINICAL TRIAL: NCT06433232
Title: Effect of Endodontic Treatment on Inflammatory Markers, Disease Activity and Periapical Healing in Rheumatoid Arthritis Patients With Apical Periodontitis : A Prospective Interventional Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Principal Investigator, Sanjay Tewari, principal pgids, Postgraduate Institute of Dental Sciences Rohtak
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bhavika Bansal
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis AND Apical Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhuematoid arhtritis patients (Experimental): Rhuematoid arhtritis patients: Change in PAI, hsCRP, ESR, SDAI and quality of life using OHIP-14 will be assessed post root canal treatment
  Interventions: Procedure: ROOT CANAL TREATMENT
- Systemically healthy patients (Active Comparator): Systemically healthy patients: Change in PAI, hsCRP, ESR, and quality of life using OHIP-14 will be assessed post root canal treatment
  Interventions: Procedure: ROOT CANAL TREATMENT

INTERVENTIONS:
Procedure: ROOT CANAL TREATMENT — ROOT CANAL TREATMENT

SUMMARY:
SUMMARY TITLE: "Effect of endodontic treatment on inflammatory markers, disease activity and periapical healing in rheumatoid arthritis patients with apical periodontitis"

RATIONALE: Chronic inflammation plays a pivotal role in rheumatoid arthritis as subjects present with elevated serum levels of numerous cytokines such as IL-1, IL-6, 1L-12, IL-17, tumour necrosis factor-alpha, RANK and RANK Ligand. Periodontal and pulpal inflammation are two major low grade chronic inflammatory diseases of the oral cavity. Apical periodontitis extends from the chronic inflammatory process that originated in the dental pulp to surround the apex of the tooth. Thus Rheumatoid arthritis and apical periodontitis converge upon common pathway of inflammation. The scientific literature has also shown to provide potential link between endodontic infection and rheumatoid arthritis. The evidence of increased prevalence of apical periodontitis in subjects of rheumatoid arthritis is provided mainly by cross-sectional and case control studies. Interventional studies have been performed in subjects with rheumatoid arthritis and periodontal disease, with results depicting beneficial effect of periodontal therapy in patients of rheumatoid arthritis. To best of our knowledge no interventional study has been performed to assess the healing pattern of apical periodontitis in subjects of rheumatoid arthritis and subsequently effect of endodontic intervention on inflammatory profile and disease burden in the same.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age of patients 30-65 years 2.Definite diagnosis of Rheumatoid arthritis based on ACR/EULAR 2010 criteria[28] i.e a score of 6 or greater out of 10 from the individual scores in four domains: number and site of involved joints (range 0-5), serological abnormality (range 0-3), elevated acute-phase response (range 0-1) and symptom duration (two levels; range 0-1) 3. The periapical index (PAI) will be used to evaluate the periapical status patients with PAI >or=3 as given by Orstavik[29] will be included 4. Presence of total teeth >/= 12

Exclusion Criteria:

1. Patients with periodontitis, pocket depth and CAL>5mm (stage 3, 4) will be excluded.
2. Pregnancy; lactation & contraceptives
3. Patients with any other systemic disease other than Rheumatoid arthritis i.e Diabetes, HIV, Chronic Liver Disease, Chronic Kidney disease and Cardiovascular disease

5. Conditions known to alter systemic inflammatory markers i.e orthopaedic trauma, surgery and viral infections 6. Patients with BMI >/= 30 7. Medications (during last 3 months) known to affect systemic inflammatory markers (systemic steroids, immunosuppressants, hormone replacement therapy, contraceptives and systemic antibiotics) 8. Smoking

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — ender matched healthy control participants to the same gender rheumatoid arthritis individuals will be analyzed.
Enrollment: 76 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in levels of hsCRP | 12 MONTHS

SECONDARY OUTCOMES:
Change in levels of ESR | 12 MONTHS
Change in SDAI | 12 MONTHS
Quality of life using OHIP-14 | 12 MONTHS

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology clinic PGIMS ROHTAK, Rohtak, India

IPD SHARING:
Plan to Share IPD: No